CLINICAL TRIAL: NCT07376772
Title: Feasibility, Preliminary Efficacy, and User Perspective Usability of Wearable Focal Vibration Therapy on Upper Extremity Function of People With Multiple Sclerosis: A Pilot Study
Brief Title: Wearable Focal Vibration Therapy on Upper Extremity Function of People With Multiple Sclerosis: A Pilot Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB202500995
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting; Upper Extremity Dysfunction
Keywords: focal vibration therapy; multiple sclerosis; upper extremity function; wearable; feasbility
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants who will recieve the focal vibration therapy
  Interventions: Device: wearable focal vibration therapy

INTERVENTIONS:
Device: wearable focal vibration therapy — The focal vibration intervention will be delivered using a modified MyoVolt wearable vibration therapy device. Each MyoVolt vibration device will be assigned to a single participant for individual use only and will be clearly labeled with a unique study ID. Devices will be distributed during the baseline training session and returned at the end of the study. To prevent unauthorized use:
  * Participants will receive training on the appropriate use and safe handling of the device.
  * Each device will be stored by the participant in their home in a designated area, along with written instructions and contact information in case of any issues.
  * The device operates only via a linked smartphone app. This will restrict unauthorized users from easily accessing or operating the device.
  * Participants will be instructed not to allow others to use the device and to report any device malfunction, loss, or suspected misuse immediately to the research team.

SUMMARY:
This pilot mixed-method study will evaluate the feasibility, preliminary efficacy, and user experience of a home-based wearable Focal Vibration Therapy (FVT) intervention for improving upper extremity (UEx) function in people with multiple sclerosis (MS). Fifteen adults with relapsing-remitting MS (PRMS) and self-reported UEx impairments will participate in a 4-week FVT program using MyovoltTM wearable FVT devices applied to arm muscles.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Confirmed diagnosis of RRMS according to the McDonald criteria (33)
* No MS relapse or exacerbation within the past 6 months (ensuring stability of symptoms)
* Self-report on clinical evidence of UEx impairment (including reduced arm/hand function, muscle weakness, spasticity, or pain).
* Stable on MS treatment for at least four weeks before recruitment, with no plans to initiate new treatments (participants may continue current treatments during the study)
* Agree and are able to use the FVT device after training.
* Sufficient proficiency in English to participate in interviews and follow instructions
* Able to visit the laboratory for assessments
* Able to provide written informed consent

Exclusion Criteria:

* Evidence of cognitive impairment that could interfere with following instructions (Mini-Montreal Cognitive Assessment score (Mini-MoCA) < 12)
* Comorbid neurological or psychiatric conditions affecting the UEx (including stroke and severe carpal tunnel syndrome) that would confound results or make FVT unsafe
* Unstable cardiac disease or any major medical illness that would preclude participation
* Any known contraindications to vibration therapy (pregnancy, acute deep vein thrombosis, severe osteoporosis, chronic migraines, epilepsy, active malignancy in the target area, unstable cardiac disease, or an implanted pacemaker without clearance)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Nine-Hole Peg Test (9HPT) | Baseline, week 4, week 8
  The Nine-Hole Peg Test (9HPT) assesses fine motor coordination and dexterity by timing how quickly participants can place and remove nine pegs from a pegboard using one hand.

SECONDARY OUTCOMES:
Arm Function in Multiple Sclerosis Questionnaire (AMSQ) | Baseline, week 4, week 8
  AMSQ is a 31-item MS-specific patient-reported outcome measure assessing arm and hand function.
Box and Block Test (BBT) | Baseline, week 4, week 8
  The Box and Block Test (BBT) measures gross motor function with high test-retest reliability by counting the number of blocks a participant can transfer over a partition from one compartment to another within 60 seconds.
Muscle Strength | Baseline, week 4, week 8
  Muscle strength will be evaluated using a handheld dynamometer. For grip strength assessment, participants will be seated with the shoulder adducted and neutrally rotated, the elbow flexed at 90 degrees, and the forearm and wrist in a neutral position. They will be instructed to squeeze the dynamometer with maximal effort for 3 seconds. Elbow flexion and extension strength will be assessed by applying the dynamometer to the distal part of the forearm as the participant resists the examiner's force for 3 seconds. The highest value from three trials in each arm and strength will be recorded and 60 seconds of recovery time will be applied between trials.
Modified Ashworth Scale (MAS) | Baseline, week 4, week 8
  The Modified Ashworth Scale (MAS) is a widely used tool that assesses spasticity by measuring resistance during passive muscle stretching, graded on a scale from 0 (no increase in muscle tone) to 4 (rigid in flexion or extension) .
Visual Analog Scale (VAS) of Pain | Baseline, week 4, week 8
  Subjective pain intensity will be measured by VAS on a scale from 0, indicating "no pain," to 10, indicating "worst possible pain". Participants will be asked about their neuropathic extremity pain in the UEx (manifesting as burning, tingling, and/or stabbing sensations), as well as pain caused by spasticity in the UEx (such as muscle stiffness or cramping). They will also be asked about instances where neuropathic pain occurs due to nonpainful stimulation such as light touch or non-extreme temperatures. Participants will rate their current UEx pain intensity, as well as the average level of UEx pain experienced over the past two weeks. Additionally, to evaluate how UEx pain has impacted their daily activities during the same period, participants will answer a modified question derived from the Chronic Pain Grade Scale.
Modified Fatigue Impact Scale (MFIS) | Baseline, week 4, week 8
  MFIS is a validated self-report questionnaire designed to evaluate the perceived impact of fatigue in people with MS. The MFIS consists of 21 items, including 9 physical, 10 cognitive, and 2 psychosocial subscale items, and assesses fatigue experienced over the past 4 weeks.
Usability | week 4, week 8
  Semi-structured interviews will be conducted with participants to explore their experiences with FVT after the post-intervention assessment and follow-up assessment. Each interview will be one-on-one, conducted by a single researcher. An open-ended interview guide will be developed to direct the conversation, covering domains of usability, acceptability, and perceived benefit of FVT.
Adherence | week 4
  Adherence to the 4-week FVT intervention will be tracked using multiple methods to ensure accuracy. Each participant will use the MyoVolt smartphone app, which automatically logs session attendance (date, time, intensity, and duration of each FVT session). The app data provides an objective record of when the device is activated. The MyoVolt app's built-in monitoring will serve as the primary source of adherence data. Participants will also fill out a simple daily adherence log immediately after each session. In this log, they will record the date and time of the session, the muscle sites stimulated (e.g., wrist extensors, biceps). This self-report acts as a cross-check against the app data and captures which muscle groups were targeted each day. Participants will be provided with a printed log template with spaces to fill in each field for every day of the 4-week intervention. This log will be collected at the post-intervention visit.
Retention rate | baseline, week 4, week 8
  Retention will be assessed by recording which participants complete the intervention and all outcome assessments. A retention log will note the status of each participant (Completed, Dropped Early, Lost to Follow-Up) and the reasons for drop-out.
Adverse events | week 4, week 8
  Participant safety will be closely monitored throughout the study. Adverse event documentation guidelines in the Agency for Healthcare Research and Quality manual were adopted. Participants will receive comprehensive information on adverse events and will be provided with diaries to record any occurrences, along with the contact information of the researcher. If an adverse event occurs, participants are instructed to immediately stop applying for FVT and contact the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwu Wang, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will collect data from a research lab and home environment. Demographics, patient-reported and clinician-performed outcome assessments on upper extremity function, and technology-based vibration dosage and usage data will be acquired from 15 participants with multiple sclerosis both in-person and remotely. Identifiable data will be de-identified prior to repository submission. The study protocol, data collection forms/case report forms, data dictionary, manual of operations, and a glossary of domain-specific terms will be submitted. Participant age, sex, ethnicity, height, weight, socioeconomic status, medication usage, upper extremity motor fuction, gross motion fuction, strength, spasticity, and pain data will be collected and shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Scientific data will be shared as soon as possible. Scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the study. The study data will be stored in the public repository for at least 5 years.
Access Criteria: Data will be stored in the UF system and sharing of de-identified data will be possible using a public repository such as the Institutional Repository at UF, as recommended by the UF Smathers Libraries Data Curation and Working Group. The study data will also be submitted to two generalist repositories participating in the NIH Generalist Repository Ecosystem Initiative, Synapse (for the wearable data) and Vivli. We will use the National Institute of Child Health and Human Development (NICHD) DASH (data and specimen hub) for repository. To promote the discoverability of the data, we will prepare a statement regarding data sharing and access to disseminate with presentations, publications, and public events related to this work. We will also submit metadata associated with the datasets to Synapse and Vivli. The repositories will provide metadata, persistent identifiers, and long-term access for open and controlled access.